CLINICAL TRIAL: NCT02133833
Title: Quantum Spectrum Radiation Emitter for Adhesive Capsulitis (Frozen Shoulder or Stiff Painful Shoulder): a Prospective, Self-controlled Trial
Brief Title: Quantum Spectrum Radiation Emitter for Adhesive Capsulitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Junxie Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 11zyy
Record Dates: First submitted 2014-03-27; First posted 2014-05-08 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quantum Spectrum Radiation Emitter (Experimental): five pieces of Quantum Spectrum Radiation Emitter will be placed on the affected shoulder daily for three weeks.
  Interventions: Device: Quantum Spectrum Radiation Emitter

INTERVENTIONS:
Device: Quantum Spectrum Radiation Emitter — The patients receive stimulation treatment of Quantum Spectrum Radiation Emitter (5 quantum chips) daily for three weeks. The emitters are placed around the shoulder.
  Other Names: Brand names: Bio-Qi

SUMMARY:
This is a prospective, self-controlled study to evaluate the efficacy of the Quantum spectrum radiation emitter for adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis (also termed frozen shoulder, stiff painful shoulder, or periarthritis) is a common cause of shoulder pain estimated to affect 2-5% of the general population.

The disorder is characterized by spontaneous onset of shoulder pain and progressive global stiffness of the glenohumeral joint accompanied by significant disability. Most studies have suggested a self-limiting condition lasting an average of two to three years, although significant numbers of people have residual clinically detectable restriction of movement beyond three years, and smaller numbers have residual disability.

Many interventions have been advocated for the treatment of adhesive capsulitis, although only limited data from randomised controlled trials are available. In addition, there are not enough data to either support or refute the efficacy of any of the commonly used interventions for this condition, including non-steroidal anti-inflammatory drugs, corticosteroid injections, and physiotherapy. Oral steroids were first advocated in the 1950s, with claims that they expedited recovery and reduced the need for manipulation under anaesthesia. However, these medications are associated with many adverse reactions.

The aims of this study are to determine whether three weeks' treatment with quantum spectrum radiation emitter in patients with adhesive capsulitis is effective for improving pain, function, and range of motion.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide written informed consent
* over 18 years old
* with pain and stiffness in one shoulder predominantly for three weeks or more
* restriction of passive motion in at least one shoulder by more than 30˚ in two or more planes of movement, measured at the time of the onset of pain with a gravity inclinometer.

Exclusion Criteria:

* hypertensive patients
* patients with cardiac arrhythmias
* patients with epilepsy
* patients with pacemakers, hearing aids or other electronic components
* pregnant patients
* patients with radiological evidence of osteoarthritis of the shoulder or fracture;calcification about the shoulder joint;reason to suspect a complete rotator cuff tear (weakness of arm elevation, a positive"drop arm sign", a high riding humerus visible on X ray of the shoulder or demonstration of a complete rotator cuff tear on ultrasound)
* patients likely not to comply with follow up (for example, living too far away to attend for follow-up assessment, or indicating they would be unable or unwilling to attend for outcome assessment)
* patients without written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
self-reported pain and function scores | at first day and 3 weeks
  Participants' overall assessment of pain, night pain, and activity related pain are each measured using a vertical Likert scale labelled"no pain"( = 0) at the bottom and"maximum imaginable pain"( = 10) at the top.
The shoulder pain and disability index | at first day and 3 weeks
  The shoulder pain and disability index (SPADI) is calculated by summing and then averaging the items of the two subscales.
Croft score | at first day and 3 weeks
  The Croft shoulder disability questionnaire are recorded as a yes or a no, and the number of positive responses is summated to give a score out of 22.
DASH score | at first day and 3 weeks
  The"disabilities arm shoulder and hand"(DASH) questionnaire has 30 items relating to functional activities and symptoms.
Participant-rated improvement | at first day and 3 weeks
  Participant-rated improvement using a five point categorical scale (marked improvement, moderate improvement, the same, moderate worsening, marked worsening).
Range of active motion | at first day and 3 weeks
  A standardised protocol is used to measure active total shoulder flexion and abduction.

SECONDARY OUTCOMES:
The health assessment questionnaire | at baseline and three weeks
  The health assessment questionnaire (HAQ) is a well validated, 9-item, arthritis specific functional assessment measure and asks about two or three fixed items in eight areas of daily life. The disability score is between 0 (no disability) and 3 (highest disability).
SF-36 | at first day and 3 weeks
  The short form 36 item health survey (SF-36) is a self administered, 36 item generic indicator of health status which consists of eight subscales representing eight dimensions of quality of life: physical function, role limitations because of physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations because of emotional problems, and general mental health. Each of the eight subscales is rescaled from 0-100; higher scores represent better health.

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Y Yuan, Principal Investigator — Nanjing Junxie Hosipital
Locations (1):
- Junxie Hospital, Nanjing, Jiangsu, China